CLINICAL TRIAL: NCT04752241
Title: Preservation of Inferior Mesenteric Artery Could Improve Sexual Function After Laparoscopic Colorectal Resection for Diverticular Disease
Acronym: IMAPSEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Saverio Mari, MD, PhD, FACS, Researcher, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DS-041
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Sexual Function Disturbances
Keywords: Sexual function; Colonic diverticular disease; Inferior mesenteric artery-preserving; Neosigmoid Denervation; Postoperative sexual dysfunction
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMAP (Experimental): Inferior Mesenteric Artery Preservation Performing left hemicolectomy and anterior rectal resection the IMA was preserved ligating close to the colonic wall the sigmoids arteries.
  Interventions: Procedure: Inferior Mesenteric Artery Preservation
- IMAS (Active Comparator): Inferior Mesenteric Artery Ligation Performing left hemicolectomy the IMA is ligated and sectioned after the origin of left colic artery
  Interventions: Procedure: Inferior Mesenteric Artery Ligation

INTERVENTIONS:
Procedure: Inferior Mesenteric Artery Preservation — Performing left hemicolectomy the IMA was preserved ligating close to the colonic wall the sigmoids arteries.
  Arms: IMAP
Procedure: Inferior Mesenteric Artery Ligation — Performing left hemicolectomy the IMA is ligated and sectioned after the origin of left colic artery
  Arms: IMAS

SUMMARY:
This study aims to evaluate whether IMA sparing may represent an advantage in terms of reduced incidence and severity of sexual dysfunctions after colorectal resections for diverticular disease (DD).

DETAILED DESCRIPTION:
Enrolled patients were randomly divided into 2 treatment groups. In the first group (IMAP) the IMA was preserved sectioning the sigmoid arteries near colonic wall while, in the second group (IMAS) the IMA was sectioned immediately below the origin of the left colic artery. Incidence and severity of sexual dysfunction and QoL were assessed by four validated questionnaire administered 6,12 months and 5 and 8 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* diverticular disease
* Diverticulitis
* BMI under 35 Kg/mq
* ASA score from I to III
* Standardized sigmoid, left colon or rectal resection

Exclusion Criteria:

* complicated diverticulitis (Hinchey III-IV)
* previous abdominal surgery or prostatic and/or gynecological resections
* adverse local condition or the need of multiorgan resection or stoma creation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Sexual disfunction 1 | 12 months after surgery
  Presence of sexual disfunction ( defined through the evaluation of sexual desire ,arousal, lubrication , orgasmic function, overall satisfaction, pain, intercourse satisfaction , erectile function)
Sexual disfunction 2 | 6 years after surgery
  Presence of sexual disfunction ( defined through the evaluation of sexual desire ,arousal, lubrication , orgasmic function, overall satisfaction, pain, intercourse satisfaction , erectile function)

SECONDARY OUTCOMES:
Sexual Function Male 1 | 12 month after surgery
  assess the patients' sexual disorders with International Index of Erectile Function (IIEF) 15-items test
Sexual Function Male 2 | 6 years after surgery
  assess the patients' sexual disorders with International Index of Erectile Function (IIEF) 15-items test
Sexual Function Female 1 | 12 months after surgery
  assess the patients' sexual disorders withFemale Sexual Function Index (FSFI) a 19-item test (score below 26.55 indicates the presence of sexual dysfunctions)
Sexual Function Female 2 | 6 years after surgery
  assess the patient's sexual disorders with Female Sexual Function Index (FSFI) 19-item test (score below 26.55 indicates the presence of sexual dysfunctions)
Quality of Life 1 | 12 months after surgery
  The impact of sexual disorders in QoL was evaluated using EORTC QLQ-30 ( European organisation for research and treatment of cancer- quality of life questionnaire)
Quality of Life 2 | 6 years after surgery
  The impact of sexual disorders in QoL was evaluated using EORTC QLQ-30( European organisation for research and treatment of cancer- quality of life questionnaire)
Quality of life SF-36 1 | 12 months after surgery
  The impact of sexual disorders in QoL was evaluated using SF-36 score (Short Form Health Survey 36)
Quality of life SF-36 2 | 6 years after surgery
  The impact of sexual disorders in QoL was evaluated using SF- 36 score ( Short Form Health Survey 36 )

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Sant'Andrea, Rome, Italy

IPD SHARING:
Plan to Share IPD: No